CLINICAL TRIAL: NCT00268229
Title: A Phase I Trial of Imatinib Mesylate (Gleevec, Formerly Known as STI571) in Combination With Daunorubicin and Cytarabine for C-kit Positive Relapsed AML
Brief Title: Imatinib Mesylate, Daunorubicin, and Cytarabine in Treating Patients With Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE-CCF-6441; P30CA043703 (NIH); CASE-CCF-6441
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute minimally differentiated myeloid leukemia (M0); adult acute megakaryoblastic leukemia (M7); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Cytarabine; Daunorubicin; Imatinib Mesylate

INTERVENTIONS:
Drug: cytarabine — 300 mg/m2/day
Drug: daunorubicin hydrochloride — 45 mg/m2/day
Drug: imatinib mesylate — dose escalation (300 mg/day to 800 mg/day).

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as daunorubicin and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving imatinib mesylate together with daunorubicin and cytarabine may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of imatinib mesylate when given together with daunorubicin and cytarabine in treating patients with relapsed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) and recommended phase II dose of imatinib mesylate in combination with daunorubicin hydrochloride and cytarabine in patients with relapsed acute myeloid leukemia.

Secondary

* Assess the non-dose-limiting toxicities associated with this regimen in these patients.
* Determine any preliminary evidence of clinical activity of this regimen in these patients.

OUTLINE: This is an open-label, dose-escalation study of imatinib mesylate.

Patients receive daunorubicin IV on days 1-3 and cytarabine IV continuously on days 1-7. Patients also receive oral imatinib mesylate once daily beginning on day 1 and continuing until disease progression or unacceptable toxicity. Patients with persistent leukemia on day 14 bone marrow biopsy but ≥ 50% reduction in bone marrow blasts receive 5 more days of cytarabine and 2 more days of daunorubicin while continuing imatinib mesylate.

Cohorts of 3-6 patients receive escalating doses of imatinib mesylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 1 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Bone marrow biopsy confirming acute myeloid leukemia (AML)

  * No M3 AML
* Patient must have relapsed to standard chemotherapy

  * Patients who relapse within six months of response to treatment or those who never responded to an anthracycline/cytarabine combination will be excluded
* At least 20% of peripheral blood or bone marrow blasts positive for c-kit
* No evidence of leptomeningeal involvement

PATIENT CHARACTERISTICS:

* ECOG Performance Status 0-2
* Liver enzymes (AST and ALT) and total bilirubin ≤ 2 times upper limit of normal
* Serum creatinine ≤ 2 times upper limit of normal
* No New York Heart Association grade III or IV cardiac problems

  * Defined as congestive heart failure or myocardial infraction within the past 6 months
* No known chronic liver disease (i.e., chronic active hepatitis and cirrhosis)
* No serious or poorly controlled medical conditions that could be exacerbated by the treatment or would seriously complicate compliance with this study
* No other active primary malignancy unless it is not currently clinically significant and does not require active intervention
* No history of HIV infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No significant history of noncompliance to medical regimens or inability to grant reliable informed consent

PRIOR CONCURRENT THERAPY:

* Previous treatment-related toxicities should be resolved
* No other investigational agents within the past 28 days
* No chemotherapy within the past 4 weeks

  * 6 weeks for nitrosourea or mitomycin C
* No major surgery within the past 4 weeks
* No concurrent use of the following drugs is allowed: ketoconazole, dilantin, itraconazole, erythromycin, clarithromycin, dexamethasone, rifampin, tegretol, phenobarbital, Hypericum perforatum (St. John's wort), cyclosporine, pimozide, warfarin, certain HMG-CoA reductase inhibitors, traizolo-benzodiazepines, or dihydropyridine calcium channel blockers
* No other concurrent anticancer agents, including chemotherapy and biologic agents
* No other concurrent investigational drugs
* Concurrent medications known to be metabolized by cytochrome p450 enzymes are allowed
* No therapeutic anticoagulation with warfarin will be permitted in patients participating in this study

  * Therapeutic anticoagulation may be accomplished using low-molecular weight heparin
  * Mini-dose warfarin for prophylaxis of central venous catheter thrombosis allowed
* No concurrent routine use of systemic corticosteroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of imatinib mesylate at one year | 1 year

SECONDARY OUTCOMES:
Non-dose limiting toxicities associated with imatinib mesylate at one year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Advani, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States